CLINICAL TRIAL: NCT01504438
Title: Prospective Randomized Evaluation Of A Two And Three Piece Total Ankle Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00031027
Record Dates: First submitted 2011-10-10; First posted 2012-01-05 (Estimated); Results first posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: Ankle Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Salto Talaris Total Ankle Replacement (Other)
  Interventions: Device: Salto-Talaris Total Ankle Replacement
- STAR Total Ankle Replacement (Other)
  Interventions: Device: STAR Total Ankle Replacement

INTERVENTIONS:
Device: Salto-Talaris Total Ankle Replacement — Salto-Talaris Total ankle replacement surgery
  Arms: Salto Talaris Total Ankle Replacement
Device: STAR Total Ankle Replacement — STAR Total Ankle Replacement
  Arms: STAR Total Ankle Replacement

SUMMARY:
This is a randomized study to prospectively compare and evaluate the functional outcome and patient satisfaction of total ankle replacements for tibio-talar osteoarthritis using either the STAR or Salto-Talaris prothesis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age > 18 years) who will benefit from a total ankle replacement, as determined by Drs. Nunley, DeOrio, or Easley, with the aid of the physical exam and routine radiography treated at Duke University Medical Center and who have no medical conditions that would represent contraindications to surgery or anesthesia will be asked to participate in this study.

Exclusion Criteria:

* The only excluded patients will be those who do not choose to participate in this study, have a weight greater than 250lbs, or do not meet the minimum age of 18 years.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A Nunley, MD, Principal Investigator — Duke University
Locations (1):
- Duke Medical Plaza Page Road, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two subjects were not randomized.
Period: Overall Study
Arm/Group | Salto-Talaris Total Ankle Replacement | STAR Total Ankle Replacement
Started | 48 | 50
Completed | 22 | 25
Not Completed | 26 | 25

BASELINE CHARACTERISTICS:
Population: Participants with data collected at all timepoints.
Groups:
- Total: Total of all reporting groups
Arm/Group | Salto-Talaris Total Ankle Replacement | STAR Total Ankle Replacement | Total
Number analyzed (Participants) | 37 | 37 | 74
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.83 (11.20) | 65.64 (8.17) | 65.73 (9.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 32 | 54
  Male | 15 | 5 | 20
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 33 | 34 | 67
  Other | 4 | 3 | 7
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37 | 37 | 74
Smoking status [Count of Participants; unit: Participants] — Population: Data not collected on 2 participants in the STAR Total Ankle Replacement group.
  Participants
    number analyzed (Participants) | 37 | 35 | 72
    Current | 2 | 0 | 2
    Former | 18 | 15 | 33
    Never | 17 | 20 | 37
Diabetes [Count of Participants; unit: Participants] — Population: Data not collected on 2 participants in the STAR Total Ankle Replacement group.
  Participants
    number analyzed (Participants) | 37 | 35 | 72
    Yes | 3 | 6 | 9
    No | 34 | 29 | 63

OUTCOME MEASURES:

1. Primary Outcome: Pain Following a Total Ankle Replacement as Measured by the Visual Analog Scale (VAS) for Pain
Description: To assess changes in pain across time following total ankle replacement. The visual analog scale (VAS) is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a mark on a 100mm line that represents a continuum between "no pain" and "worst pain." A score of 0 represents less pain intensity while a score of 100 represents high pain intensity
Time Frame: Baseline, 6 months, 1 year, 2 years, 3 years
Population: Data not collected at 3 years.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- STAR: STAR Total Ankle Replacement
Arm/Group | Salto-Talaris Total Ankle Replacement | STAR
Number analyzed (Participants) | 37 | 37
mm
  Baseline: number analyzed (Participants) | 35 | 36
  Baseline | 67.0 (25.9) | 71.3 (21.4)
  6 months: number analyzed (Participants) | 34 | 36
  6 months | 16.7 (22.9) | 18.6 (20.0)
  1 year: number analyzed (Participants) | 35 | 37
  1 year | 12.0 (19.1) | 16.9 (20.8)
  2 years: number analyzed (Participants) | 29 | 33
  2 years | 12.4 (19.4) | 23.5 (28.7)
  3 years: number analyzed (Participants) | 0 | 0
Statistical Analysis 1: Comparison: Salto-Talaris Total Ankle Replacement vs STAR; Test type: Other; p = 0.29, ANOVA

2. Primary Outcome: Functional Health Following a Total Ankle Replacement Using the 36-Item Short Form Health Survey (SF-36).
Description: The SF-36 comprises 36 questions which cover eight domains of health: Limitations in physical activities because of health problems, Limitations in social activities because of physical or emotional problems, Limitations in usual role activities because of physical health problems, Bodily pain, General mental health (psychological distress and well-being), Limitations in usual role activities because of emotional problems, Vitality (energy and fatigue), and General health perceptions. Scores for the different domains are converted and pooled using a scoring key, for a total score indicating a range of low to high Quality of Life (QOL). Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability
Time Frame: Baseline, 6 months, 1 year, 2 years, 3 years
Population: Data not collected at 3 years.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Salto-Talaris Total Ankle Replacement | STAR Total Ankle Replacement
Number analyzed (Participants) | 37 | 37
score on a scale
  Baseline: number analyzed (Participants) | 33 | 34
  Baseline | 69.1 (19.3) | 67.4 (22.1)
  6 months: number analyzed (Participants) | 31 | 32
  6 months | 47.7 (17.4) | 51.4 (19.1)
  1 year: number analyzed (Participants) | 31 | 33
  1 year | 71.4 (18.7) | 70.7 (21.2)
  2 years: number analyzed (Participants) | 27 | 31
  2 years | 77.1 (17.3) | 69.5 (21.6)
  3 years: number analyzed (Participants) | 0 | 0
Statistical Analysis 1: Comparison: Salto-Talaris Total Ankle Replacement vs STAR Total Ankle Replacement; Test type: Other; p = 0.31, ANOVA

3. Primary Outcome: Physical Limitations Following a Total Ankle Replacement as Measured by the Short Musculoskeletal Function Assessment (SMFA) Questionnaire.
Description: The SMFA consists of two sections: 34 questions covering the assessment of the patient's function and 12 questions covering how bothered patients are by their symptoms. Items are scored in six categories: daily activities, emotional status, arm and hand function, mobility category, and bother index. On a scale of 1 to 5, patients rate their ability on each item and higher total scores represent greater degree of dysfunction or bother. SMFA higher total score represent greater degree of dysfunction or bother. The lowest score is 0 representing the best possible function and the highest score is 100 representing an overall higher degree of dysfunction or bother.
Time Frame: Baseline, 6 months, 1 year, 2 years, 3 years
Population: Data not collected at 3 years.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Salto-Talaris Total Ankle Replacement | STAR Total Ankle Replacement
Number analyzed (Participants) | 37 | 37
score on a scale
  Baseline: number analyzed (Participants) | 35 | 36
  Baseline | 83.0 (19.2) | 80.3 (19.5)
  6 months: number analyzed (Participants) | 34 | 36
  6 months | 54.9 (14.7) | 60.4 (18.7)
  1 year: number analyzed (Participants) | 35 | 37
  1 year | 51.5 (12.6) | 57.1 (15.6)
  2 years: number analyzed (Participants) | 29 | 34
  2 years | 48.5 (12.9) | 56.1 (18.9)
  3 years: number analyzed (Participants) | 0 | 0
Statistical Analysis 1: Comparison: Salto-Talaris Total Ankle Replacement vs STAR Total Ankle Replacement; Test type: Other; p = 0.07, ANOVA

4. Primary Outcome: Pain and Function Following a Total Ankle Replacement as Measured by the American Orthopaedic Foot and Ankle Society (AOFAS) Ankle-Hindfoot Rating System
Description: The AOFAS Ankle-Hindfoot Rating System is a standardized evaluation of the clinical status of the ankle-hindfoot. Patients report their pain and physicians assess alignment; the patient and physician work together to complete the functional portion. Scores range from 0 to 100, with healthy ankles receiving 100 points.
Time Frame: Baseline, 6 months, 1 year, 2 years, 3 years
Population: Data not collected at 3 years.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Salto-Talaris Total Ankle Replacement | STAR Total Ankle Replacement
Number analyzed (Participants) | 37 | 37
score on a scale
  Baseline: number analyzed (Participants) | 31 | 32
  Baseline | 44.6 (14.9) | 46.4 (17.9)
  6 months: number analyzed (Participants) | 29 | 28
  6 months | 80.2 (13.5) | 76.1 (17.3)
  1 year: number analyzed (Participants) | 27 | 24
  1 year | 84.5 (9.9) | 78.0 (12.9)
  2 years: number analyzed (Participants) | 21 | 24
  2 years | 84.5 (9.3) | 64.7 (23.7)
  3 years: number analyzed (Participants) | 0 | 0
Statistical Analysis 1: Comparison: Salto-Talaris Total Ankle Replacement vs STAR Total Ankle Replacement; Test type: Other; p = 0.04, ANOVA

5. Primary Outcome: To Measure a Change in One's Daily Activity Following a Total Ankle Replacement Using the Foot and Ankle Disability Index (FADI) at Multiple Time Points.
Description: The FADI has 26 items, each of which is scored from 0 (unable to do) to 4 (no difficulty at all). The four pain items of the FADI are scored 0 (none) to 4 (unbearable). The total score ranges 0 to 104 with higher scores indicating a better outcome.
Time Frame: Baseline, 6 months, 1 year, 2 years, 3 years
Population: Data not collected at 3 years.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Salto-Talaris Total Ankle Replacement | STAR Total Ankle Replacement
Number analyzed (Participants) | 37 | 37
score on a scale
  Baseline: number analyzed (Participants) | 26 | 21
  Baseline | 55.1 (18.9) | 51.6 (13.3)
  6 months: number analyzed (Participants) | 2 | 2
  6 months | 8.0 (11.3) | 51.5 (17.7)
  1 year: number analyzed (Participants) | 15 | 11
  1 year | 20.1 (21.5) | 26.2 (13.7)
  2 years: number analyzed (Participants) | 6 | 10
  2 years | 16.0 (15.1) | 18.0 (18.7)
  3 years: number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Three Dimensional Kinematic and Kinetic Assessment During Level Walking Across Time Following Total Ankle Replacement.
Description: In order to understand the effect of the ankle replacement on lower extremity kinematics and kinetics, each subject will be asked to complete a series of functional tasks and level walking trials at each of the study timepoints.
Time Frame: Baseline, 6 months, 1 year, 2 years, 3 years
Population: Data not collected.
Arm/Group | Salto-Talaris Total Ankle Replacement | STAR Total Ankle Replacement
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 7 years
Arm/Group | Salto-Talaris Total Ankle Replacement | STAR Total Ankle Replacement
All-Cause Mortality (participants affected / at risk) | 0/48 | 1/50
Serious Adverse Events (participants affected / at risk) | 0/48 | 1/50
Other Adverse Events (participants affected / at risk) | 0/48 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Salto-Talaris Total Ankle Replacement (N=48) | STAR Total Ankle Replacement (N=50)
Death (General disorders) | 0 | 1 — Unrelated to study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-12-15): https://cdn.clinicaltrials.gov/large-docs/38/NCT01504438/Prot_SAP_000.pdf